CLINICAL TRIAL: NCT06353997
Title: A Phase II, Single-arm, Multi-center, Open-label Study of Neoadjuvant INBRX-106 (Hexavalent OX40 Agonist) in Combination With Pembrolizumab as an Induction Immunotherapy for Stage II/III TNBC Patients
Brief Title: Neoadjuvant INBRX-106 in Combination With Pembrolizumab for Stage II/III TNBC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Inhibrx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024000099
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + INBRX-106 (Experimental): Patients will be given pembrolizumab at a dose of 200mg IV in combination with INBRX-106 at a dose of 0.1mg/kg IV every 3 weeks.
  Interventions: Drug: Pembrolizumab; Drug: INBRX-106

INTERVENTIONS:
Drug: Pembrolizumab — Drug will be delivered per standard-of-care as established by trial Keynote-522.
  Other Names: KEYTRUDA
Drug: INBRX-106 — INBRX-106 is a hexavalent, recombinant humanized IgG1, OX40 agonist antibody that targets the human OX40 receptor (TNFRSF4, UniProtKB: P43489). INBRX-106 is based on a sdAb platform and, in detail, 3 identical humanized camelid heavy chain-only antibody binding domains (VHHs) targeting OX40 are joined end-to-end and with an Fc based on human IgG1 to create a molecule that homo-dimerizes into an antibody targeting a total of 6 OX40 receptors.

SUMMARY:
This is a Phase II trial to assess efficacy and feasibility of pembrolizumab + INBRX-106 as an induction therapy preceding neoadjuvant therapy.

DETAILED DESCRIPTION:
A Simon 2-stage design is implemented to minimize exposure if the treatment regimen is not feasible or if no response. If feasibility is established with responses exceeding futility parameters, study will expand to stage 2. Additional arms may be introduced in a protocol amendment.

Below shows the sample size required using Simon's 2-stage design, 80% power and 5% one-sided significance level:

* Null hypothesis: <5% week 6 US response
* Alternative hypothesis: >35% week 6 US response
* Stage I n (r*): 6 (0)
* Stage I + II total n (r): 12 (2)
* Criteria: Minimax
* Minimum responses to proceed to stage II: 1

Note: r* and r represents the threshold for declaring futility, i.e. greater than r* or r responses would be required to consider ongoing investigation.

The null hypothesis of 5% is based upon the assumption that virtually no subjects would experience volumetric reduction if the therapy was not effective. The alternative hypothesis of 35% is based upon the assumption that responses in the absence of chemotherapy in approximately one-third of subjects would be clinically meaningful, encouraging further development of the treatment paradigm.

If no responses are observed, a second feasibility run-in may be considered using a biomarker enrichment strategy (such as with the 27-gene IO score).

The arm will be terminated from further development if an unacceptable proportion of patients experience rapid clinical/radiographic progression (defined as progression of disease, or clinical evidence of progression), or other toxicities that interfere with curative-intent therapy, defined as >1/6 evaluable subjects in stage I or >2/12 in stage II, evaluated for each arm. This is a Pocock-type stopping boundary that yields the probability of cross the boundary at most 23% when the rate of dose-limiting toxicity is equal to 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, inclusive of all genders.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 2.
3. Patients must have histologically confirmed TNBC (ER/PR ≤ 10% allowed, HER2- as defined by ASCO guidelines). HER2 negative permitted to enroll as IHC 0, 1, or 2+ with negative ISH.
4. Primary breast tumor measurable by ultrasound and at least 1cm.
5. Clinically appropriate to receive neoadjuvant pembrolizumab plus chemotherapy (e.g. Keynote-522) planned for curative intent per standard of care (as indicated following study therapy however not mandated on trial for Option 2).
6. Multifocal/multicentric disease is allowed. If clinically indicated per the standard of care, suspicious sites that do not appear to be part of the same disease process should be biopsied with reconfirmation of ER/PR/HER2 status. Up to 20 slides or 1 block may be submitted to conduct biomarkers studies on remaining tissue.
7. No prior therapy of any kind for TNBC.
8. Willingness to undergo serial ultrasounds, serial biopsies, and blood draws.
9. Patients must have adequate organ function as defined below. Specimens must be collected within 28 days prior to the start of study treatment.

   * Absolute neutrophil count (ANC) ≥1500/µL
   * Platelets ≥100 000/µL
   * Hemoglobin ≥8.0 g/dL or ≥5.0 mmol/L
   * Creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
   * Total bilirubin ≤1.5 × ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN. Patients with elevated LFTs that are suggestive of Gilbert's disease (a benign process) are eligible.
   * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN
   * International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
   * TSH and free T4 levels should be drawn within 14 days prior to start of treatment. Patients must have adequate thyroid function as demonstrated by free T4 values, regardless of TSH.
10. Fertile male patients and female patients of childbearing potential must agree to avoid impregnating a partner or becoming pregnant, respectively. They must be willing to employ highly effective contraception methods (with a failure rate of less than 1% when used consistently and correctly) at least 28 days before the first dose of study treatment until 4 months after the last dose of study treatment.

    A woman is considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. Postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

    Acceptable methods of contraception presented below are in compliance with the Clinical Trial Facilitation and Coordination Group (CTFG) recommendations related to contraception and pregnancy testing in clinical trials, Version 1.1 (September, 2020). However, if a contraception method listed below is restricted by local regulations/guidelines, then it does not qualify as an acceptable method of contraception in that country/region. Local guidelines should be followed.
    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: Oral. Intravaginal. Transdermal.
    * Progestogen-only hormonal contraception associated with inhibition of ovulation: Oral. Injectable. Implantable.
    * Intrauterine device (IUD).
    * Intrauterine hormone-releasing system (IUS).
    * Bilateral tubal occlusion.
    * Vasectomized partner. (Only considered to be highly effective contraception if he is the sole sexual partner of the female patient of childbearing potential and if the vasectomized partner has received medical assessment of the surgical success.)
    * Sexual abstinence. (Only considered to be highly effective contraception if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient and if considered acceptable by local regulatory agencies and IRBs/IECs.
11. WOCBP must have a negative urinary or serum pregnancy test within 72 hours prior to start of treatment. If screening serum pregnancy test collected outside of 72 hours prior to start of treatment, this may be accepted for determination of eligibility but must be re-checked prior to treatment C1D1. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The following age-specific requirements apply:

    Women < 50 years of age are considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

    Women ≥ 50 years of age are considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
12. To be eligible by H&E, the tumor must have a stromal tumor infiltrating lymphocytes (sTILs) score of at least 1% on diagnostic biopsy as defined by the International TILs Working Group (https://www.tilsinbreastcancer.org/), ascertained by local pathologist or study pathologist.

Exclusion Criteria:

1. Bilateral breast cancer.
2. Prior malignancies that require ongoing active therapy or are at clinically significant risk of systemic recurrence in the opinion of the investigator.
3. Suspicion for, or histologically confirmed, metastatic disease.
4. Primary tumor with potential for skin ulceration or invasion of the chest wall, or with pain that would suggest rapid progression or imminent muscle/skin involvement in the opinion of the enrolling investigator.
5. Prior therapy with an anti-PD-1, anti-PD-L1, or antiPDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137). Patients who have received these agents more than 3 years prior for other malignancies may be considered if they are not still at clinically significant risk of systemic recurrence in the opinion of the investigator.
6. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
7. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

   Additionally, COVID-19 vaccinations (including boosters) should not be scheduled within 72 hours (before or after) of dosing days for INBRX-106 and pembrolizumab.
9. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
10. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Pregnant or breastfeeding.
12. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. History of allogenic tissue/solid organ transplantation.
14. Has active autoimmune disease that has required systemic treatment in excess of prednisone 10mg daily or equivalent in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Has a known additional malignancy (other than their current breast cancer diagnosis) that is progressing or has required active systemic treatment within the past 3 years.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
15. History or current evidence of any condition, therapy, or clinically significant laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Active infection requiring systemic therapy with the exception of UTI requiring oral antibiotic therapy and prophylactic anti-viral therapy (e.g. Acyclovir).
17. Known history of Human Immunodeficiency Virus (HIV) infection.
18. Known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Patients with naturally acquired immunity are allowed (i.e. HBsAg(-); HBcAb(+); HBsAb(+/-).
19. Any known history of active TB (Bacillus Tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Volumetric Response | At the end of Cycle 2 (each cycle is 21 days)
  Patients achieving (>30%) reduction in ultrasound estimate of breast mass volume (mL) at the end of 2 cycles investigational therapy

SECONDARY OUTCOMES:
Pathological response (following extended INBRX-106 + pembrolizumab) | 30 days from last dose of study treatment
  Patients achieving pathological response after completion of study therapy followed by additional neoadjuvant therapy per treating physician discretion, ascertained at the time of definitive surgery.
Pathological response (post-chemotherapy) | 30 days from last dose of study treatment
  Number of patients achieving pathological response following extended anti-OX40 + pembrolizumab if continued beyond 2 cycles (option 2).
IO-path response assessed prior to Cycle 2 | Day 21
  On study biopsy conducted prior to Cycle 2:
  * IO-path-NE (not evaluable): no tumor or evidence of treatment effect.
  * IO-path-NR (no response): tumor present, no appreciable treatment effect, no sTILs/iTILs expansion by at least 10% absolute increase from baseline.
  * IO-path-PR (partial response): tumor present, +treatment effect and/or sTILs/iTILs expansion by at least 10% absolute increase from baseline.
  * IO-path-CR (complete response): no viable tumor, + treatment effect.
Event free survival | Up to 2 years
  Date of dose 1 until evidence of cancer recurrence or death. Those alive without recurrence are censored at 5 years after the last dose of study drug.
Overall survival | Up to 2 years
  Date of dose 1 to death. Those who are alive are censored at 5 years after the last dose of study drug.
Toxicity profile | 30 days from last dose of study treatment
  All AEs attributed to study therapy per CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: David Page, MD, Principal Investigator — Providence Health & Services
Locations (4):
- United States (4):
  - Ellison Institute of Technology (EITM), Los Angeles, California
  - Providence Portland Cancer Institute - Franz Clinic, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Swedish Cancer Institute, Seattle, Washington